CLINICAL TRIAL: NCT01869998
Title: Implication of Left veNtricle Vortex Flow Guided aNticOagulation Therapy for preVenting Apical Thrombus Formation In Patients With Acute myOcardial infarctioN: Multicenter Prospective Randomized Clinical Trial; INNOVATION Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0040
Record Dates: First submitted 2013-05-30; First posted 2013-06-05 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Apical Thrombus Formation; Acute Myocardial Infarction
Keywords: Vortex; Thrombus; Contrast echocardiography; Prediction and prevention of apical thrombus formation in acute myocardial infarction patient by using Vortex parameters.
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Low risk group (A): (A)Vortex depth≥0.45
- High risk group 1 (B): (B)Vortex depth<0.45 with anticoagulation
- High risk group 2 (C): (C)Vortex depth <0.45 without anticoagulation

SUMMARY:
Implication of left veNtricle vortex flow guided aNticOagulation therapy for preVenting Apical Thrombus formation In patients with acute myOcardial infarctioN: Multicenter Prospective Randomized Clinical Trial; INNOVATION study

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 30 years old
2. Acute anterior wall myocardial infarction showing akinetic or dyskinetic apical wall motion abnormalities on an initial transthoracic echocardiogram
3. Left ventricular ejection fraction less than 40%

Exclusion Criteria:

1. Prior history of myocardial infarction
2. Chronic medication with Coumadin
3. Contraindication of contrast echocardiography
4. Significant atrial or ventricular arrhythmia
5. Valvular heart disease more than moderate degree
6. Decompensated heart failure
7. Very poor echo window, which cannot evaluate the presence of apical thrombus

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute anterior wall myocardial infarction showing akinetic or dyskinetic apical wall motion abnormalities on an initial transthoracic echocardiogram
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Apical thrombus formation in echocardiography | 30 days after initial echocardiography
  Evaluate and compare the incidence of thrombus formation in high risk group (Vortex depth < 0.45) and low risk group (Vortex Depth ≥ 0.45)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance cardiovascular hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Son JW, Park WJ, Choi JH, Houle H, Vannan MA, Hong GR, Chung N. Abnormal left ventricular vortex flow patterns in association with left ventricular apical thrombus formation in patients with anterior myocardial infarction: a quantitative analysis by contrast echocardiography. Circ J. 2012;76(11):2640-6. doi: 10.1253/circj.cj-12-0360. Epub 2012 Aug 7. PMID 22878352